CLINICAL TRIAL: NCT02823522
Title: Non-Celiac Wheat Sensitivity: Permanent or Transient Condition? A Follow-up Study
Brief Title: Non-Celiac Wheat Sensitivity: Permanent or Transient Condition?
Status: Recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Other Study IDs: ACPM11
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Non-Celiac Wheat Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patients recruitment — Between July and November 2016, the patients included in the previous retrospective study were contacted by phone, mail and e-mail and invited to come back to the respective clinics where they had been initially diagnosed as NCWS patients: the Department of Internal Medicine of the University Hospital of Palermo and the Department of Internal Medicine of the Hospital of Sciacca (province of Agrigento).

SUMMARY:
Non-Celiac Gluten Sensitivity (NCGS) has been recently included among the gluten-related diseases. Patients suffering from NCGS are diagnosed after carefully excluding celiac disease (CD), and immunoglobulin E (IgE)-mediated wheat allergy. Then, in the absence of sensitive and specific diagnostic biomarkers for NCGS, a monitoring of the patient during elimination and re-introduction of wheat by a double-blind placebo controlled (DBPC) challenge method has been suggested as diagnostic hallmark. Some studies seem to suggest that wheat components other than gluten can cause the symptoms, and therefore the term "non-celiac wheat sensitivity" (NCWS) has been proposed instead of NCGS. While it is well known that CD is a long-life condition and a strict adherence to the gluten-free diet must be maintained, it is unknown whether this is valid for NCWS. On the year 2012, the researchers published a retrospective study, including 276 patients with irritable bowel syndrome (IBS)-like symptoms who had been diagnosed with NCWS using a DBPC challenge during a ten-years period (2001-2011). The present prospective study aimed to evaluate: A) how many of these patients are still following a wheat-free diet, and B) which percentage was still suffering from NCWS, diagnosed by DBPC wheat challenge, in a subgroup of that cohort.

DETAILED DESCRIPTION:
Non-Celiac Gluten Sensitivity (NCGS) has been recently included among the gluten-related diseases. Patients suffering from NCGS are diagnosed after carefully excluding celiac disease (CD) diagnosis by negative CD-specific serum antibodies and absence of intestinal villi atrophy, and excluding IgE-mediated wheat allergy, by negative serum specific IgE and/or skin prick test with wheat antigens. Then, in the absence of sensitive and specific diagnostic biomarkers for NCGS, a monitoring of the patient during elimination and re-introduction of wheat by a double-blind placebo controlled (DBPC) challenge method has been suggested as diagnostic hallmark. Obviously, this a cumbersome and time-consuming procedure which has been used in few studies.

Despite an increasing percentage of the general population define themselves as "gluten-sensitive", and by the year 2017 the market of the gluten-free products will be worth 6.6 billion of dollars, doubts persist about many aspects of NCGS. Some studies seem to suggest that wheat components other than gluten can cause the symptoms, and therefore the term "non-celiac wheat sensitivity" (NCWS) has been proposed instead of NCGS. Furthermore, while it is well known that CD is a long-life condition and a strict adherence to the gluten-free diet must be maintained, it is unknown whether this is valid for NCWS.

On the year 2012, the researchers published a retrospective study, including 276 patients with irritable bowel syndrome (IBS)-like symptoms who had been diagnosed with NCWS using a DBPC challenge during a ten-years period (2001-2011).

The present prospective study aimed to evaluate the persistence of the NCWS condition in that cohort and, consequently, the researchers estimated : A) how many of these patients are still following a wheat-free diet, and B) which percentage was still suffering from NCWS, diagnosed by DBPC wheat challenge, in a subgroup of that cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with NCWS by DBPC challenge.

Exclusion Criteria:

* The 22 patients, included in the previous study, who tested positives for anti-endomysial antibodies (EmA) in the culture medium of the duodenal biopsies, even if the villi/crypts ratio in the duodenal mucosa was normal, were excluded from the present study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the previous retrospective study were contacted by phone, mail and e-mail and invited to come back to the respective clinics where they had been initially diagnosed as NCWS patients: the Department of Internal Medicine of the University Hospital of Palermo and the Department of Internal Medicine of the Hospital of Sciacca.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2024-08 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
How many patients were still following a gluten-free or a wheat-free diet | Between July and November 2016
  A structured questionnaire was administered to evaluate how many patients were still following a gluten-free diet (GFD) and how many a wheat-free diet.

SECONDARY OUTCOMES:
Evaluation of the effect of the GFD on IBS symptoms | Between July and November 2016
  The researchers administered a modified version of the IBS Global Assessment of Improvement (IBS-GAI) score. A responder was defined as a patient whose symptoms were either 'moderately improved' or 'substantially improved' compared with the period preceding the NCWS diagnosis.
Evaluation of the severity of the IBS condition | Between July and November 2016
  The researchers administered the IBS Symptom Severity Scale (IBS-SSS), evaluating the change in total IBS-SSS score from the first evaluation (time of the NCWS diagnosis) and the follow-up evaluation (present study). A respondent was classified as a patient whose overall symptom severity on the IBS-SSS changed >50 points.
Re-evaluation of the NCWS condition by DBPC-Wheat challenge | Between July and November 2016
  Finally, the repetition of the DBPC-wheat challenge will be proposed to the patients still on GFD. Those who will accept will be randomized to undergo the challenge. It will be performed with the same method used in the retrospective study.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Principal Investigator — Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sapone A, Bai JC, Ciacci C, Dolinsek J, Green PH, Hadjivassiliou M, Kaukinen K, Rostami K, Sanders DS, Schumann M, Ullrich R, Villalta D, Volta U, Catassi C, Fasano A. Spectrum of gluten-related disorders: consensus on new nomenclature and classification. BMC Med. 2012 Feb 7;10:13. doi: 10.1186/1741-7015-10-13. PMID 22313950
- [Background] Ludvigsson JF, Leffler DA, Bai JC, Biagi F, Fasano A, Green PH, Hadjivassiliou M, Kaukinen K, Kelly CP, Leonard JN, Lundin KE, Murray JA, Sanders DS, Walker MM, Zingone F, Ciacci C. The Oslo definitions for coeliac disease and related terms. Gut. 2013 Jan;62(1):43-52. doi: 10.1136/gutjnl-2011-301346. Epub 2012 Feb 16. PMID 22345659
- [Background] Catassi C, Elli L, Bonaz B, Bouma G, Carroccio A, Castillejo G, Cellier C, Cristofori F, de Magistris L, Dolinsek J, Dieterich W, Francavilla R, Hadjivassiliou M, Holtmeier W, Korner U, Leffler DA, Lundin KE, Mazzarella G, Mulder CJ, Pellegrini N, Rostami K, Sanders D, Skodje GI, Schuppan D, Ullrich R, Volta U, Williams M, Zevallos VF, Zopf Y, Fasano A. Diagnosis of Non-Celiac Gluten Sensitivity (NCGS): The Salerno Experts' Criteria. Nutrients. 2015 Jun 18;7(6):4966-77. doi: 10.3390/nu7064966. PMID 26096570
- [Background] Spence D. Bad medicine: food intolerance. BMJ. 2013 Jan 30;346:f529. doi: 10.1136/bmj.f529. No abstract available. PMID 23364064
- [Background] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Background] Fasano A, Sapone A, Zevallos V, Schuppan D. Nonceliac gluten sensitivity. Gastroenterology. 2015 May;148(6):1195-204. doi: 10.1053/j.gastro.2014.12.049. Epub 2015 Jan 9. PMID 25583468
- [Background] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Derived] Carroccio A, D'Alcamo A, Iacono G, Soresi M, Iacobucci R, Arini A, Geraci G, Fayer F, Cavataio F, La Blasca F, Florena AM, Mansueto P. Persistence of Nonceliac Wheat Sensitivity, Based on Long-term Follow-up. Gastroenterology. 2017 Jul;153(1):56-58.e3. doi: 10.1053/j.gastro.2017.03.034. Epub 2017 Mar 30. PMID 28365444